CLINICAL TRIAL: NCT05448729
Title: Shear Wave Elastography Versus Strain Elastography With Histogram Analysis in Solid Pancreatic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Dr. Seicean Andrada, Professor, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 396/2022
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Endoscopic Ultrasonography
Keywords: elastography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strain ratio Elastography EUS (Sham Comparator): The solid pancreatic lesion will be assessed by using strain ratio elastography EUS
  Interventions: Diagnostic Test: Elastography EUS
- Shear Wave Elastography EUS (Active Comparator): The solid pancreatic lesion will be assessed by using shear wave elastography EUS
  Interventions: Diagnostic Test: Elastography EUS

INTERVENTIONS:
Diagnostic Test: Elastography EUS — Comparison between the values of strain ratio and shear wave in concordance with the final diagnosis

SUMMARY:
to assess the diagnostic value of strain elastography EUS and shear wave EUS in solid pancreatic lesions

DETAILED DESCRIPTION:
Three measurements of strain ratio elastography and three measurements of shear wave elastography with VPN> 20% will be performed in the same solid pancreatic lesions. The results will be compared in the groups of adenocarcinomas, neuroendocrine tumors and benign solid pancreatic lesions.

ELIGIBILITY:
Inclusion Criteria:

* patients with solid pancreatic masses > 2 cm in diameter at CT scan for EUS assessment

Exclusion Criteria:

* Patients with inconclusive pathology results
* patients with cystic component > 20%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity | 12 months
  Comparison between the diagnostic rate in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Andrada Seicean, Prof, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy Cluj-Napoca

IPD SHARING:
Plan to Share IPD: Yes
Patients inclusions in another medical center
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12 luni
Access Criteria: Web connection

REFERENCES:
- [Result] Ohno E, Kawashima H, Ishikawa T, Iida T, Suzuki H, Uetsuki K, Yashika J, Yamada K, Yoshikawa M, Gibo N, Aoki T, Kataoka K, Mori H, Yamamura T, Furukawa K, Nakamura M, Hirooka Y, Fujishiro M. Diagnostic performance of endoscopic ultrasonography-guided elastography for solid pancreatic lesions: Shear-wave measurements versus strain elastography with histogram analysis. Dig Endosc. 2021 May;33(4):629-638. doi: 10.1111/den.13791. Epub 2020 Sep 15. PMID 32662150
- See also: DOI: 10.1111/den.13791 — https://pubmed.ncbi.nlm.nih.gov/32662150/